CLINICAL TRIAL: NCT06867250
Title: Evaluation of Peri-Implant Sulcus Fluid Vitamin D and Cathelicidin (LL-37) Levels in Peri-Implant Health and Diseases
Brief Title: Peri-implant Vitamin D and Cathelicidin (LL-37) Levels
Status: Completed | Type: Observational
Sponsor: Altinbas University (Other)
Responsible Party: Principal Investigator, ILKNUR OZENCI, Assistant professor, Altinbas University
Other Study IDs: 2021/45
Record Dates: First submitted 2025-03-03; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Peri-Implantitis and Peri-implant Mucositis
Keywords: peri-implant sulcus fluid; peri-implant diseases; LL-37; 25(OH)D
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Peri-implant sulcus fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- peri-implant healthy, peri-implant mucositis, peri-implantitis: A total of 105 dental implants from 33 patients were assessed, with 35 categorized in the peri-implant health group, 35 in the peri-implant mucositis group, and 35 in the peri-implantitis group.
  Interventions: Diagnostic Test: The patients' periodontal clinical parameters were recorded. PISF samples were collected, and the evaluations of 25(OH)D and LL-37 were conducted using enzyme-linked immunosorbent assay.

INTERVENTIONS:
Diagnostic Test: The patients' periodontal clinical parameters were recorded. PISF samples were collected, and the evaluations of 25(OH)D and LL-37 were conducted using enzyme-linked immunosorbent assay. — In vitro studies have shown that vitamin D promotes the release of antimicrobial peptides from gingival epithelial cells, no clinical research has specifically examined its effect on LL-37 levels in peri-implant tissue diseases. This study seeks to investigate the relationship between vitamin D levels in peri-implant sulcus fluid and clinical parameters in individuals with both peri-implant health and disease. Additionally, it aims to assess the correlation between vitamin D and the antimicrobial peptide LL-37.

SUMMARY:
This research aims to explore the influence of vitamin D on the body's defense system by examining its impact on specific proteins involved in immune response and inflammation in the soft tissues surrounding dental implants. Also aims to determine how vitamin D levels affect these proteins and their role in protecting peri-implant tissues from microbial infections and inflammation.

DETAILED DESCRIPTION:
This cross-sectional clinical study examined 33 patients with 105 dental implants, classified as having either healthy peri-implant tissues or peri-implant diseases. Participants had not received peri-implant treatment in the past six months or taken medications affecting peri-implant tissues in the last three months. Eligible implants had been functional for at least 12 months with prosthetic superstructures that allowed sample collection. Patients with uncontrolled systemic conditions, metabolic bone diseases, autoimmune disorders, or those who were pregnant or breastfeeding were excluded.

Clinical assessments were conducted at six peri-implant sites, measuring probing depth (PD), clinical attachment level (CAL), modified plaque index (mPI), modified sulcus bleeding index (mSBI), and keratinized mucosa width (KMW). Bone loss was evaluated using radiographs. Patients were categorized into three groups based on the 2017 Classification of Periodontal and Peri-implant Diseases: peri-implant health, peri-implant mucositis, and peri-implantitis (35 implants per group).

Peri-implant sulcus fluid (PISF) samples were collected for 25(OH)D and LL-37 analysis using enzyme-linked immunosorbent assay (ELISA). Statistical analysis included normality tests (Kolmogorov-Smirnov), descriptive statistics, one-way ANOVA with Tukey HSD, Kruskal-Wallis with Dunn's test, chi-square tests, and Spearman's correlation for non-normally distributed data.

ELIGIBILITY:
Inclusion Criteria:

* Not received peri-implant treatment in the previous six months.
* Had not used vitamin D supplements, antibiotics, anti-inflammatory drugs, or any medications that could affect peri-implant tissues in the last three months.
* Patients with dental implants had been in function for at least 12 months, had been under functional loading for at least six months, and had prosthetic superstructures that allowed for unobstructed sample collection.

Exclusion Criteria:

* Uncontrolled systemic conditions, disorders affecting peri-implant tissues, metabolic bone diseases, autoimmune disorders.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This cross-sectional clinical study included 33 patients with dental implants, exhibiting either healthy peri-implant tissues or peri-implant diseases, who sought treatment at the Department of Periodontology, Faculty of Dentistry, Altınbaş University.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Peri-implant sulcus fluid vitamin D levels and clinical parameters correlation | At the day of visit (Day 0)- Peri-implant clinical assessments and peri-implant sulcus fluid collection
  The association between vitamin D levels in peri-implant sulcus fluid and clinical parameters in individuals with peri-implant health and peri-implant diseases.
The correlation between vitamin D and the antimicrobial peptide LL-37 | Laboratory tests were completed after all samples were collected.
  Peri-implant sulcus fluid Vitamin d and LL-37 levels were investigated with ELISA
Mucosal Inflammation | At the day of visit (Day 0)
  Measurement of mucosal inflammation around implants using modified plaque index (mPI), and modified sulcus bleeding index (mSBI).
Probing Pocket Depth | At the day of visit (Day 0)
  Measurement of the periodontal pockets depth around implants. Unit of Measure: Millimeters (mm)
Width of Keratinized Mucosa | At the day of visit (Day 0)
  Measurement of the width of keratinized mucosa around the implants. Unit of Measure: Millimeters (mm)

CONTACTS AND LOCATIONS:
Overall Officials: ILKNUR OZENCI, Dr, Principal Investigator — Altinbas University
Locations (1):
- Altinbas University, Istanbul, BAKIRKOy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This detailed description provides a comprehensive overview of your study, outlining its objectives, background, methodology, and expected outcomes in a structured and academic manner.